CLINICAL TRIAL: NCT02966301
Title: Phase II Study of First Line Treatment of Chronic Graft Versus Host Disease With Arsenic Trioxide
Brief Title: Treatment of Chronic Graft Versus Host Disease With Arsenic Trioxide
Acronym: GvHD-ATO
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Medsenic (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GMED16-001
Record Dates: First submitted 2016-10-28; First posted 2016-11-17 (Estimated); Results first posted 2022-05-09 (Actual); Last update posted 2022-05-09 (Actual); Status verified 2020-07

CONDITIONS: Chronic Graft-Versus-Host Disease; Immune System Diseases
Keywords: cGvHD; Arsenic Trioxide; Hematology
MeSH Terms: conditions — Bronchiolitis Obliterans Syndrome; Immune System Diseases | interventions — Arsenic Trioxide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- interventional (Experimental): Single arm : Arsenic trioxide
  Interventions: Drug: Arsenic Trioxide Injectable Solution

INTERVENTIONS:
Drug: Arsenic Trioxide Injectable Solution — Each patient will receive eleven perfusions of arsenic trioxide (0,15 mg/kg/Day - IV administration) over a 4 weeks period (one cycle).
  Patients in partial response after the 1st cycle of ATO will be eligible to receive a second cycle of ATO as consolidation therapy. A delay of 8 weeks (from the first infusion of ATO) will be observed between the two cycles of ATO therapy.
  The study duration will be 2 years (12 months recruitment + 12 months follow-up).
  Other Names: Trisenox / Arscimed

SUMMARY:
This study aims to evaluate the early chronic GvHD events (first line therapy), if the addition of arsenic trioxide to standard therapy with corticosteroids, with or without cyclosporine, will be effective in controlling chronic GvHD and to reduce the duration of corticosteroid therapy

DETAILED DESCRIPTION:
Graft-versus-host disease (GvHD) is the most common long-term complication in patients who underwent allogeneic transplantation.

First-line therapy for chronic GVHD is based on immunosuppressive agents (corticosteroids with or without cyclosporine) achieving satisfactory response in around 30% of patients.

This is a prospective, national, multicenter, non-randomized Phase II study that will include a total number of 24 patients in which, trioxide d'arsenic will be administrated at 0,15mg/kg/day.

Clinical response will be evaluated based on the Working Group Report 2015, published by the National Institute of Health Consensus.

Follow-up visits will be weekly for four weeks (ATO cycle), every two weeks from second to third month of ATO treatment, every month from the fourth to sixth month of ATO treatment and every 3 months, at 9 months and 12 months (final visit).

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (≥18 years) who have received a first allogeneic stem cell transplantation for a hematological disease (any source of hematopoietic stem cells is authorized; any category of conditioning regimen prior to allo-SCT is authorized; any type of stem cell donors is authorized)
* Confirmed diagnosis of a first episode of chronic GvHD requiring systemic immunosuppressive therapy (any prior GvHD prophylaxis previously used is accepted). Chronic GvHD diagnosis is defined according to the NIH Working Group Consensus. Chronic GvHD diagnosis will be based on the evaluation of the severity of the different clinical manifestations including:

  * Performance status evaluation
  * Cutaneous evaluation measured by the percentage of extension or the presence of sclerotic features. If relevant, confirmation with a biopsy should be performed whenever possible
  * Oral symptoms
  * Ocular symptoms
  * Gastro-intestinal symptoms
  * Evaluation of liver involvement (total bilirubin, transaminases and alkaline phosphatases)
  * Pulmonary function evaluation
  * Evaluation of the musculoskeletal manifestations, especially the amplitude of the relevant articulations
  * Genital tract symptoms
* Signed informed consent
* Absence of contra-indications to the use of ATO
* Subjects affiliated with an appropriate social security system
* Men must use a medically acceptable method of contraception throughout the treatment period and for at least 4 months and 10 days following the last treatment administration
* Women who are of childbearing potential must have a negative serum pregnancy test and agree to use a medically acceptable method of contraception throughout the study and for 3 months following the end of the study
* Patient not participating or not having participated in a clinical study in the 30 days prior to his/her inclusion in the study

Exclusion Criteria:

* Patient developing acute GvHD (whether early or "late onset" form)
* Patients developing overlap GvHD as defined by the 2014 NIH Working Group Consensus (presence of one or more acute GvHD manifestations in a patient with a diagnosis of chronic GvHD)
* A "mild" form of chronic GvHD not requiring systemic immunosuppressive therapy
* A "moderate" form of chronic GvHD limited to one organ site not requiring systemic immunosuppressive therapy
* Patient receiving mycophenolate mofetil
* Not the first episode of chronic GvHD needing systemic immunosuppressive therapy
* Second allogeneic stem cell transplant
* Severe cardiac diseases (congestive heart failure (NYHA class III), recent myocardial infarction (in the past 6 months before the inclusion), histories of unexplained syncope, ...)
* Significant arrhythmias, electrocardiogram (EKG) abnormalities:
* Congenital QT syndromes
* History or presence of significant ventricular or atrial tachyarrhythmia
* Clinically significant resting bradycardia (< 50 beats per minutes)
* QTc>450msecformenand>470msecfor women on screening EKG (using the QTcF formula)
* Right bundle branch block plus left anterior hemiblock, bifascicular block
* Central or peripheral neuropathy
* Neutrophils < 0.5 × 109/L
* Platelets < 50 × 109/L
* Potassium ≤ 4 mEq/l*
* Magnesium ≤ 1.8 mg/dl*
* Calcium ≤ 2.15 mmol/l*
* Hepatic impairment due to a suspected or proven liver damage, other than direct hepatic cGvHD involvement
* PT < 50%
* Renal impairment (creatinine ≥ 100 μmol/l)
* Uncontrolled systemic infection which in the opinion of the investigator is associated with an increased risk of the patients' death within 1 month after the start of therapy
* Severe neurological or psychiatric disorders
* Denied informed consent
* Pregnancy
* Women breastfeeding at selection and throughout the treatment period

  * If abnormal at selection, to be corrected and re-validated following electrolytes infusion, before inclusion and each drug perfusion.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2016-12 (Actual); Primary Completion 2020-06 (Actual); Study Completion 2020-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mohamad Mohty, Pr, Principal Investigator — Hôpital Saint-Antoine, AP-HP - Paris; Anne Huyhn, Dr, Principal Investigator — Institut Universitaire du Cancer - Oncopole - Toulouse; Sylvain Chantepie, Dr, Principal Investigator — Institut d'Hématologie de Basse Normandie - CHU de Caen; Patrice Chevallier, Dr, Principal Investigator — Hôtel Dieu - CHU Nantes; Didier Blaise, Pr, Principal Investigator — Institut Paoli Calmettes - Centre de Recherche en Cancérologie de Marseille; Patrice Ceballos, Dr, Principal Investigator — Hôpital St Eloi - Montpellier; Patrice Turlure, Dr, Principal Investigator — University Hospital, Limoges; Edouard Forcade, Dr, Principal Investigator — University Hospital, Bordeaux

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Rongvaux-Gaida D, Dupuis M, Poupon J, Djebrani-Oussedik N, Lemonnier C, Rieger F. High Response Rate and Corticosteroid Sparing with Arsenic Trioxide-Based First-Line Therapy in Chronic Graft-versus-Host Disease after Allogeneic Hematopoietic Stem Cell Transplantation. Transplant Cell Ther. 2022 Oct;28(10):679.e1-679.e11. doi: 10.1016/j.jtct.2022.07.004. Epub 2022 Jul 10. PMID 35830931

RESULTS

PARTICIPANT FLOW:
Groups:
- Arsenic Trioxide Injectable Solution: Single arm : Arsenic trioxide Injectable Solution
  Arsenic Trioxide Injectable Solution: Each patient will receive eleven perfusions of arsenic trioxide (0,15 mg/kg/Day - IV administration) over a 4 weeks period (one cycle).
  Patients in partial response after the 1st cycle of ATO will be eligible to receive a second cycle of ATO as consolidation therapy. A delay of 8 weeks (from the first infusion of ATO) will be observed between the two cycles of ATO therapy.
  The study duration will be 2 years (12 months recruitment + 12 months follow-up).
Period: Overall Study
Arm/Group | Arsenic Trioxide Injectable Solution
Started | 21
Full Analysis Set (FAS) | 20 (All patients who entered the study, completed their first cycle of ATO (11 infusions) and for whom the response at Week 6 after diagnosis of chronic GvHD has been evaluated.)
Safety Analysis (SA) | 21 (All patients included in the study for whom received at least one ATO infusion. One patient received 2 infusions and then exited the study due to SAE (reversible liver toxicity).)
Completed | 18
Not Completed | 3
Not completed — Death | 2
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Groups:
- Arsenic Trioxide: Single arm : Arsenic trioxide
  Each patient will receive eleven perfusions of arsenic trioxide (0,15 mg/kg/Day - IV administration) over a 4 weeks period (one cycle).
  Patients in partial response after the 1st cycle of ATO will be eligible to receive a second cycle of ATO as consolidation therapy. A delay of 8-10 weeks (from the first infusion of ATO) will be observed between the two cycles of ATO therapy.
  The study duration was 3.5 years (36 months recruitment + 12 months follow-up).
Arm/Group | Arsenic Trioxide
Number analyzed (Participants) | 21
Age, Continuous [Mean (Full Range); unit: years] | 62 [42 to 72]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11
  Male | 10
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  France | 21
Diagnosis of chronic GvHD requiring systemic immunosuppressive therapy confirmed, [Count of Participants; unit: Participants] — Only patients meeting the National Institutes of Health (NIH) criteria for chronic GvHD requiring systemic therapy were eligible for inclusion in this study
  Participants | 21

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Complete or Partial Remission of Chronic Graft Versus Host Disease After a First Line Treatment With Arsenic Trioxide
Description: Clinical response will be evaluated based on the Working Group Report 2015, published by the National Institute of Health Consensus.
  Response definition is as follows:
  * Complete remission (CR) is defined as complete disappearance of any sign of chronic GvHD.
  * Partial remission (PR) is defined as a significant improvement as defined by the organ or site specific measurement scale without progression in any other organ or site.
Time Frame: six months
Population: All patients who entered the study, completed their first cycle of ATO and for whom the response at Week 6 after diagnosis of chronic GvHD has been evaluated.
Measure: Count of Participants; unit: Participants
Groups:
- Interventional: Single arm : Arsenic trioxide Injectable Solution
  Arsenic Trioxide Injectable Solution: Each patient will receive eleven perfusions of arsenic trioxide (0,15 mg/kg/Day - IV administration) over a 4 weeks period (one cycle).
  Patients in partial response after the 1st cycle of ATO will be eligible to receive a second cycle of ATO as consolidation therapy. A delay of 8 weeks (from the first infusion of ATO) will be observed between the two cycles of ATO therapy.
  The study duration will be 2 years (12 months recruitment + 12 months follow-up).
Arm/Group | Interventional
Number analyzed (Participants) | 20
Participants | 15

2. Secondary Outcome: Average Dose of Corticosteroids
Description: Average dose in mg/kg/day of prednisone or prednisone equivalent
Time Frame: Average dose of Prednisone at 6 months after the first infusion of ATO
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mg/kg/day
Arm/Group | Interventional
Number analyzed (Participants) | 20
mg/kg/day | 0.22 (0.29)

3. Secondary Outcome: Failure Free Survival
Description: Treatment failure were defined by:
  * Initiation of a new systemic treatment for chronic GvHD;
  * Recurrent or progressive malignancy;
  * Death
Time Frame: 6 months after first ATO infusion
Population: FAS
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Interventional
Number analyzed (Participants) | 20
percentage of participants | 90 [65.6 to 97.4]

4. Secondary Outcome: Number of Adverse Events
Description: Tolerability and safety of ATO in combination with Prednisone, with or without Ciclosporine, in patients with chronic GvHD after allo-SCT.
  Adverse events follow-up for all patients throughout the study
Time Frame: 12 months after the first infusion of ATO for each patient
Population: Safety Analysis Population
Measure: Number; unit: number of events
Arm/Group | Interventional
Number analyzed (Participants) | 21
number of events | 197

5. Secondary Outcome: Cumulative Incidence for Non-relapse Mortality (NRM)
Description: Non-Relapse Mortality (NRM) of infectious and non-infectious origin
Time Frame: 12 months after first ATO infusion
Population: FAS
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Interventional
Number analyzed (Participants) | 20
percentage of participants | 5 [0.3 to 21.1]

ADVERSE EVENTS:
Time Frame: For each patient the specific period over which data on adverse events were collected is 1 year after inclusion in the clinical study
Groups:
- Arsenic Trioxide Infusion: Single arm : Arsenic trioxide Injectable Solution
Arm/Group | Arsenic Trioxide Infusion
All-Cause Mortality (participants affected / at risk) | 2/21
Serious Adverse Events (participants affected / at risk) | 21/21
Other Adverse Events (participants affected / at risk) | 21/21
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arsenic Trioxide Infusion (N=21)
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Respiratory tract infection viral (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pancytopenia (Blood and lymphatic system disorders) | 1 (1)
Encephalopathy (Nervous system disorders) | 1 (1)
Epilepsy (Nervous system disorders) | 1 (1)
Oedema peripheral (General disorders) | 1 (1)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1)
Hepatitis acute (Hepatobiliary disorders) | 1 (1)
Hepatotoxicity (Hepatobiliary disorders) | 2 (2)
Septic shock (Infections and infestations) | 1 (1)
Urinary tract infection (Infections and infestations) | 3 (3)
Genital herpes (Infections and infestations) | 1 (1)
Oropharyngeal candidiasis (Infections and infestations) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1)
Sepsis (Infections and infestations) | 1 (1)
Escherichia pyelonephritis (Infections and infestations) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arsenic Trioxide Infusion (N=21)
Hyperaemia (Vascular disorders) | 1 (2)
Hypertension (Vascular disorders) | 1 (1)
Thrombosis (Vascular disorders) | 1 (1)
Venous thrombosis (Vascular disorders) | 1 (1)
Drug hypersensitivity (Immune system disorders) | 1 (1)
Hypogammaglobulinaemia (Immune system disorders) | 2 (2)
Asthenia (General disorders) | 3 (3)
Chest pain (General disorders) | 1 (1)
Cyst (General disorders) | 1 (1)
Face oedema (General disorders) | 1 (1)
Influenza like illness (General disorders) | 1 (1)
Medical device pain (General disorders) | 1 (1)
Mucosal inflammation (General disorders) | 1 (1)
Oedema peripheral (General disorders) | 7 (8)
Pain (General disorders) | 1 (1)
Pyrexia (General disorders) | 5 (7)
Insomnia (Psychiatric disorders) | 2 (2)
Irritability (Psychiatric disorders) | 1 (1)
Sleep disorder (Psychiatric disorders) | 1 (1)
Vulvovaginal dryness (Reproductive system and breast disorders) | 2 (2)
Vulvovaginal erythema (Reproductive system and breast disorders) | 1 (1)
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 1 (1)
Scar (Injury, poisoning and procedural complications) | 1 (1)
Blood lactate dehydrogenase increased (Investigations) | 1 (1)
Cardiac murmur (Investigations) | 1 (1)
CD4 lymphocytes decreased (Investigations) | 1 (2)
Electrocardiogram QT prolonged (Investigations) | 1 (1)
Angina pectoris (Cardiac disorders) | 2 (2)
Atrial fibrillation (Cardiac disorders) | 2 (2)
Cough (Respiratory, thoracic and mediastinal disorders) | 9 (10)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Obstructive airways disorder (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pulmonary mass (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Rales (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Anaemia (Blood and lymphatic system disorders) | 2 (2)
Thrombocytopenia (Blood and lymphatic system disorders) | 2 (2)
Dizziness (Nervous system disorders) | 1 (1)
Dysgeusia (Nervous system disorders) | 1 (1)
Headache (Nervous system disorders) | 1 (1)
Paraesthesia (Nervous system disorders) | 1 (1)
Peroneal nerve palsy (Nervous system disorders) | 1 (1)
Seizure (Nervous system disorders) | 1 (1)
Dry eye (Eye disorders) | 1 (1)
Keratitis (Eye disorders) | 1 (1)
Ocular discomfort (Eye disorders) | 1 (2)
Vision blurred (Eye disorders) | 1 (1)
Visual acuity reduced (Eye disorders) | 1 (1)
Vertigo (Ear and labyrinth disorders) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 3 (4)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 8 (10)
Dysphagia (Gastrointestinal disorders) | 1 (1)
Haemorrhoids (Gastrointestinal disorders) | 1 (1)
Mouth haemorrhage (Gastrointestinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 2 (2)
Odynophagia (Gastrointestinal disorders) | 1 (1)
Rectal haemorrhage (Gastrointestinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1)
Hepatocellular injury (Hepatobiliary disorders) | 2 (4)
Dermatitis exfoliative generalised (Skin and subcutaneous tissue disorders) | 1 (1)
Eczema (Skin and subcutaneous tissue disorders) | 1 (1)
Erythema (Skin and subcutaneous tissue disorders) | 3 (3)
Ingrowing nail (Skin and subcutaneous tissue disorders) | 1 (1)
Lichenification (Skin and subcutaneous tissue disorders) | 1 (1)
Nail bed bleeding (Skin and subcutaneous tissue disorders) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (2)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (3)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 2 (2)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1)
Cushing's syndrome (Endocrine disorders) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 2 (2)
Fluid retention (Metabolism and nutrition disorders) | 1 (1)
Hyperkalaemia (Metabolism and nutrition disorders) | 2 (2)
Hypocalcaemia (Metabolism and nutrition disorders) | 1 (1)
Hypokalaemia (Metabolism and nutrition disorders) | 4 (5)
Hypomagnesaemia (Metabolism and nutrition disorders) | 2 (2)
Malnutrition (Metabolism and nutrition disorders) | 1 (1)
Bronchitis (Infections and infestations) | 1 (1)
Campylobacter infection (Infections and infestations) | 1 (1)
Conjunctivitis (Infections and infestations) | 2 (2)
Cytomegalovirus infection (Infections and infestations) | 2 (3)
Device related infection (Infections and infestations) | 2 (2)
Epstein-Barr virus infection (Infections and infestations) | 1 (1)
Escherichia urinary tract infection (Infections and infestations) | 2 (2)
Fungal infection (Infections and infestations) | 1 (1)
Genital herpes (Infections and infestations) | 1 (1)
Genital infection fungal (Infections and infestations) | 1 (1)
Klebsiella infection (Infections and infestations) | 1 (1)
Oral herpes (Infections and infestations) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1)
Pseudomonal bacteraemia (Infections and infestations) | 1 (1)
Respiratory syncytial virus infection (Infections and infestations) | 1 (1)
Rhinovirus infection (Infections and infestations) | 1 (1)
Staphylococcal infection (Infections and infestations) | 1 (1)
Staphylococcal sepsis (Infections and infestations) | 1 (1)
Urinary tract infection (Infections and infestations) | 2 (7)
Viral infection (Infections and infestations) | 1 (1)
Vulvovaginal mycotic infection (Infections and infestations) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2018-12-18): https://cdn.clinicaltrials.gov/large-docs/01/NCT02966301/Prot_000.pdf
  • Statistical Analysis Plan (2020-12-21): https://cdn.clinicaltrials.gov/large-docs/01/NCT02966301/SAP_001.pdf